CLINICAL TRIAL: NCT01441557
Title: Pilot Study on the Usefulness of 3,4-diaminopyridine in the Treatment of Botulism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI11-PR-DUPONT
Record Dates: First submitted 2011-09-26; First posted 2011-09-27 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Botulism
Keywords: mechanical ventilation
MeSH Terms: conditions — Botulism | interventions — Amifampridine

INTERVENTIONS:
Drug: 3,4-diaminopyridine — test dose 10 mg then 20 mg, then depending on tolerance and efficacy full-dose administration(from 10mg /8h to 20 mg /8h)

SUMMARY:
Main objectives:

Evaluate the effectiveness of an administration of 3,4-diaminopyridine (FIRDAPSE ®) in severe botulinic poisoning in measuring the effect on electrophysiological and respiratory parameters

Secondary Objective:

Study the natural history of electrophysiological and respiratory parameters during the botulinic intoxication

Primary endpoint:

Clinical, electrophysiological and respiratory before and after administration of 3,4-diaminopyridine.

Study Design:

Pilot study, prospective, interventional.

Study population:

Case series (n = 8 patients) suffering from botulinic type A, respiratory failure, but with no other organ failure

Experimental treatment :

3,4-diaminopyridine, FIRDAPSE ® (BioMarin) The dosage will be gradually increased according to a predetermined scheme and will not exceed 60 mg / day and 20 mg / dose.

Statistics:

Intra-individual comparison of physiological parameters measured before and after administration of 3,4-diaminopyridine. Electromyographic and respiratory parameters will be measured for each patient. Then a dose of 10 mg of 3,4-diaminopyridine will be administrated. If this dose is well tolerated and provides a relative improvement of 10% for at least one of the parameters studied, the dose will be maintained at 10 mg for 48 hours 3 times a day then increased to 20 mg.

The primary endpoint is the change in the amplitude of muscle response evaluated by the subtraction of amplitude at T1.5 and T0.

DETAILED DESCRIPTION:
Main objectives:

Evaluate the effectiveness of an administration of 3,4-diaminopyridine (FIRDAPSE ®) in severe botulinic poisoning in measuring the effect on electrophysiological and respiratory parameters

Secondary Objective:

Study the natural history of electrophysiological and respiratory parameters during the botulinic intoxication

Primary endpoint:

Clinical, electrophysiological and respiratory before and after administration of 3,4-diaminopyridine.

Study Design:

Pilot study, prospective, interventional.

Study population:

Case series (n = 8 patients) suffering from botulinic type A, respiratory failure, but with no other organ failure

Experimental treatment :

3,4-diaminopyridine, FIRDAPSE ® (BioMarin) The dosage will be gradually increased according to a predetermined scheme and will not exceed 60 mg / day and 20 mg / dose.

Statistics:

Intra-individual comparison of physiological parameters measured before and after administration of 3,4-diaminopyridine. Electromyographic and respiratory parameters will be measured for each patient. Then a dose of 10 mg of 3,4-diaminopyridine will be administrated. If this dose is well tolerated and provides a relative improvement of 10% for at least one of the parameters studied, the dose will be maintained at 10 mg for 48 hours 3 times a day then increased to 20 mg.

The primary endpoint is the change in the amplitude of muscle response evaluated by the subtraction of amplitude at T1.5 and T0.

Quantitative variables are expressed as mean ± standard deviation or median (minimum - maximum) and qualitative variables as percentages.

The null hypothesis (the evolution is identical between the two doses) will be rejected in favour of the alternative hypothesis (the evolution is different) using the mixed model analysis of variance on the threshold of 5% for the first kind with adjusting the amplitude at T0, age, the time between patient admission and the first administration of 3,4-diaminopyridine. The evolution of latency and respiratory parameters will be analyzed with the same mixed ANOVA without risk adjustment alpha.

For the secondary objective, the evolution curves of the amplitude of muscle response on the one hand and respiratory function on the other hand, will be built for each patient.

The mean (or median) of amplitude and respiratory function at weaning will be calculated with a confidence level of 95% (or range). The average time between the first 3,4-diaminopyridine administration and withdrawal of mechanical ventilation will also be calculated.

For each dose, the average evolution of the amplitude will be calculated with a confidence level of 95%.

Statistical analysis will be carried out using SAS software version 9.2.

ELIGIBILITY:
Inclusion Criteria:

* botulism
* ventilation

Exclusion Criteria:

* renal failure
* cardiac failure
* pregnancy
* under age 18
* hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
electrophysiological | 90 min
  Primary endpoint:
  Clinical, electrophysiological and respiratory before and after administration of 3,4-diaminopyridine.

CONTACTS AND LOCATIONS:
Overall Officials: Herve DUPONT, Md, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU, Amiens, France

REFERENCES:
- [Result] Friggeri A, Marcon F, Marciniak S, Lemaire-Hurtel AS, Seydi A, Ammenouche N, Levrard M, Mahjoub Y, Airapetian N, Tinturier F, Petitjean M, Dupont H. 3,4-Diaminopyridine may improve neuromuscular block during botulism. Crit Care. 2013 Sep 5;17(5):449. doi: 10.1186/cc12880. No abstract available. PMID 24007658